CLINICAL TRIAL: NCT06327347
Title: Comparative Study of 2 Multifocal Intraocular Lenses in Heidelberg
Acronym: C2H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cristalens Industrie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-05_C2H
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Lens Implantation, Intraocular; Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Parallel Assignement
Who Masked: Outcomes Assessor
Masking Description: The Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) assessed at 80 cm in photopic conditions at minimum 1-month post-operative is perforemd by a blinded evaluator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARTIS SYMBIOSE (Active Comparator): 25 patients will be implanted bilaterally with Artis Symbiose IOLs (Cristalens Industrie, France) . The device is CE-marked and used according to the intended purpose.
  Interventions: Device: intraocular lens implantation in cataract surgery
- PANOPTIX (Active Comparator): 25 patients will be implanted bilaterally with AcrySof IQ PanOptix IOLs (Alcon, Switzerland).The device is CE-marked and used according to the intended purpose.
  Interventions: Device: intraocular lens implantation in cataract surgery

INTERVENTIONS:
Device: intraocular lens implantation in cataract surgery — Implantation of intra ocular lenses in both patient's eyes in remplacement of the natural cataracted cristallin that has been removed from the patient's eye during the cataract surgery

SUMMARY:
The goal of this clinical trial is to compare the performance of 2 intraocular lenses (IOLs): ARTIS SYMBIOSE (study lenses) vs PANOPTIX (comparator) through binocular Distance Corrected Intermediate Visual Acuity (DCIVA) assessed at 80 cm in photopic conditions at minimum 1-month post-operative by a blinded evaluator.

This main objective will be to show superiority of the ARTIS SYMBIOSE system on the primary endpoint.

The patient population to be included is patient suffering from cataract who requires cataract surgery procedure that meet the inclusion and non-inclusion criteria and provide written informed consent.

Participants will attend a total of 5 study visits: 1 preoperative visit, 1 surgery visit and 3 postoperative visits.

DETAILED DESCRIPTION:
This trial is a single center, prospective, randomized (1:1), unblinded, controlled study conducted in Germany according to Art. 82 MDR (PMCF study).

The lead investigator at the Heidelberg Eye University Hospital - International Vision Correction Research Centre (IVCRC) is Pr. Gerd Auffarth.

This study examines the visual performance of the two IOLs involved : Artis Symbiose (study lenses) compared to PanOptix (comparator) in bilaterally implanted patients.

The aim of this comparative study is to assess the performance and safety of these two IOLs with targeting to demonstrate the superiority of Artis Symbiose in some specific performance parameters. The tested hypothesis is the superiority of Artis Symbiose over PanOptix IOLs on the primary evaluation criterion.

A total of 50 patients will be included at one investigational center. Subjects participating in the study will attend a maximum of 5 study visits (1 preoperative, 1 operative and 3 postoperative visits) over a period of 12 months.

Only patients who have age-related cataracts will be included in the study. To participate in this study, patients must be at least 50 years old at the time of screening and maximum 85 years old. All patients who would like to take part in this study will receive a detailed study information by the investigator staff and a written informed form. Before a patient is admitted, he or she must sign a consent form.

The primary study endpoint is to compare the performance of 2 IOLs (Artis Symbiose, and PanOptix) through Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) assessed at 80 cm in photopic conditions at minimum 1-month post-operative by a blinded evaluator.

The entire study including data processing will be carried out in accordance with EN ISO 14155:2020 Clinical Investigation of Medical Devices for Human Subjects, EN ISO 11979-7:2018: Clinical investigations of intraocular lenses for the correction of aphakia, EU MDR 2017/745, MEDDEV 2.7.1 rev. 4 Clinical Evaluation: A Guide for Manufacturers and Notified Bodies, MPDG:2020: Medical Device Law Implementation Act, as well as applicable local regulations and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 50 < Age < 85 years old
* Bilateral age-related cataract
* Signed informed consent of the study
* Availability, willingness and sufficient cognitive awareness to comply with study procedures
* No previous refractive or ocular surgery
* Need for IOL in this diopter range: 10 to 30 D
* Expected postoperative astigmatism ≤ 0.75 D
* Eye dryness ≤ 2 in dry eye severity grading
* For women of childbearing potential: Willing to adhere to an adequate form of contraception.

Non-inclusion criteria :

* Being under guardianship / curatorship
* Illiterate or not enough knowledge of German language
* Acute or chronic disease or illness that would increase risk or confound study results found to be relevant by the investigators
* Pupil > 4mm or < 2mm in photopic conditions
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* Occupation requiring night-time driving or any occupation incompatible with multifocality
* Amblyopia, strabismus, color blindness
* Extremely shallow anterior chamber
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, uveitis, Marfan's syndrome)
* Irregular astigmatism, unstable cornea
* Pregnant or women of childbearing potential or breastfeeding women

Exclusion Criteria:

* Patient consent withdrawal
* Inability to place the intraocular lens safely at the location planned.
* Surgical complications (e.g. non-circular rhexis, oversized or undersized rhexis). Each patient with these intraoperative complications should not be implanted with the study IOL.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Binocular Distance Corrected Intermediate Visual Acuity | one month
  The primary endpoint is Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) assessed at 80 cm in photopic conditions minimum 1-month post-operative by a blinded evaluator

CONTACTS AND LOCATIONS:
Locations (1):
- Universitäts-Augenklinik Heidelberg International Vision Correction Research Centre (IVCRC), Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No